CLINICAL TRIAL: NCT05143905
Title: A Phase I Randomised Single-blind Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7503 Following Single Ascending Dose Administration to Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7503 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D9230C00001
Record Dates: First submitted 2021-11-23; First posted 2021-12-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Healthy Participants
Keywords: First-in-Human; Placebo-controlled; AZD7503; Single Ascending Dose; Sentinel Dosing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: This study is single blind with regard to treatment (AZD7503 or placebo). This means that the participant and the study centre staff will remain blinded during the dosing phase of the study and the randomisation code will only be available at each pre defined decision point before the Safety Review Committee meeting in order to review the data unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1: AZD7503 dose 1 (Experimental): Randomised healthy participants will receive a single dose 1 of AZD7503.
  Interventions: Drug: AZD7503
- Cohort 2: AZD7503 dose 2 (Experimental): Randomised healthy participants will receive a single dose 2 of AZD7503.
  Interventions: Drug: AZD7503
- Cohort 3: AZD7503 dose 3 (Experimental): Randomised healthy participants will receive a single dose 3 of AZD7503.
  Interventions: Drug: AZD7503
- Cohort 4: AZD7503 dose 4 (Experimental): Randomised healthy participants will receive a single dose 4 of AZD7503.
  Interventions: Drug: AZD7503
- Cohort 5 : AZD7503 dose X (Experimental): Randomised healthy participants will receive a single dose X of AZD7503.
  Interventions: Drug: AZD7503
- Cohort 6: AZD7503 dose Y (Experimental): Randomised healthy participants will receive a single dose Y of AZD7503.
  Interventions: Drug: AZD7503
- Pooled Placebo for AZD7503 (Cohorts 1 to 6) (Placebo Comparator): Randomised healthy participants will receive placebo.
  Interventions: Drug: Placebo
- Japanese Cohort 1: AZD7503 dose 3 (Experimental): Randomised healthy Japanese participants will receive a single dose 3 of AZD7503.
  Interventions: Drug: AZD7503
- Japanese Cohort 2: AZD7503 dose 4 (Experimental): Randomised healthy Japanese participants will receive a single dose 4 of AZD7503.
  Interventions: Drug: AZD7503
- Placebo (Japanese Cohorts) (Placebo Comparator): Randomised healthy Japanese participants will receive placebo.
  Interventions: Drug: Placebo
- Chinese Cohort: AZD7503 dose 4 (Experimental): Randomised healthy Chinese participants will receive a single dose 4 of AZD7503.
  Interventions: Drug: AZD7503
- Placebo (Chinese Cohort) (Placebo Comparator): Randomised healthy Chinese participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7503 — Randomised participants will receive a single ascending dose of AZD7503 by SC injection (dose 1, dose 2, dose 3, dose 4, dose X and dose Y).
  Arms: Chinese Cohort: AZD7503 dose 4; Cohort 1: AZD7503 dose 1; Cohort 2: AZD7503 dose 2; Cohort 3: AZD7503 dose 3; Cohort 4: AZD7503 dose 4; Cohort 5 : AZD7503 dose X; Cohort 6: AZD7503 dose Y; Japanese Cohort 1: AZD7503 dose 3; Japanese Cohort 2: AZD7503 dose 4
Drug: Placebo — Randomised participants will receive placebo by SC injection
  Arms: Placebo (Chinese Cohort); Placebo (Japanese Cohorts); Pooled Placebo for AZD7503 (Cohorts 1 to 6)

SUMMARY:
This study will evaluate safety, tolerability and pharmacokinetics (PK) of AZD7503, following subcutaneous (SC) administration of single ascending doses of AZD7503 in healthy participants.

DETAILED DESCRIPTION:
This is a Phase I, First-in-Human, study in healthy males and females (non-childbearing potential) participants. In this study up to four dose levels of AZD7503 are planned to be evaluated.

The planned doses of AZD7503 are dose 1, dose 2, dose 3, and dose 4. Eligible participants will be randomised to receive either AZD7503 or placebo. The study will include four single dose cohorts with an option to include two cohorts based on emerging data from planned cohorts in the study and two additional cohorts of Japanese participants and one cohort of Chinese participants will also be included.

Dosing for each ascending dose cohort will be proceeded with sentinel dosing strategy. Here, sentinel sub-cohort will be included, such that 1 participant will be randomised to receive placebo and 1 participant will be randomised to receive AZD7503. The safety data from the sentinel participants up to 24 hours post-dose will be reviewed by the Principal Investigator (PI) before the remaining participants in the cohort are dosed

The study will comprise:

* A Screening Period of maximum 28 days;
* A Treatment Period during which participants will be resident at the Study Centre from the day before study medication administration (Day -1) until at least 72 hours after study medication administration; discharged from the Study Centre on Day 4;
* Follow-up Visits on 1,2,4,6 and 8 weeks; and
* A Final Follow-up Visit 10 weeks after the last study medication dose. Each participant will be involved in the study for approximately 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non smoking male and/or female (of non childbearing potential) participants with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the study centre, must not be lactating and must be of non childbearing potential.
* Body mass index (BMI) between 18 and 30 kg/m^2, inclusive, and weigh at least 60 kg for healthy participants or between 18 and 32 kg/m^2, inclusive, and weigh at least 50 kg for Japanese and Chinese participants.
* For Japanese and Chinese participants:

  1. A Japanese participant is defined as having both parents and 4 grandparents who are ethnically Japanese. This includes first-, second-and third-generation Japanese whose parents or grandparents are living in a country other than Japan.
  2. A Chinese participant is defined as having both parents and 4 grandparents who are ethnically Chinese. This includes first-, second-and third-generation Chinese whose parents or grandparents are living in a country other than China.
* Willing to participate in retrospective genotyping analysis for HSD17B13.

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of administration of study intervention.
* Any laboratory values with the following deviations at screening and/or Day 1:

  * Alanine aminotransferase > Upper Limit of Normal (ULN)
  * Aspartate aminotransferase > ULN
  * Total bilirubin > ULN
  * Creatinine > ULN
  * White blood cell count < Lower Limit of Normal (LLN)
  * Hemoglobin < LLN
  * Estimated glomerular filtration rate < 60 mL/min/1.73 m^2
  * Platelets >ULN and/or <LLN.
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results other than those described above, including participants with platelet or bleeding disorders, known platelet dysfunction disorders.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody or Human Immunodeficiency Virus.
* Confirmed coronavirus disease 2019 (COVID-19) infection during screening and/or admission by polymerase chain reaction (PCR) test.
* Abnormal vital signs, after 5 minutes supine rest
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the previous 3 months.
* History of alcohol abuse or excessive intake of alcohol
* History of Drug abuse or positive screen for drug of abuse or cotinine (nicotine) or alcohol.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7503.
* Excessive intake of caffeine containing drinks or food (eg, coffee, tea, chocolate)
* Use of any prescribed or non prescribed medication during the 2 weeks prior to the administration of study intervention or longer if the medication has a long half-life.
* Plasma donation within one month of screening or any blood donation/blood loss more than 500 mL during the 3 months prior to screening.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days (or 5 half lives, whichever is longer) of the administration of study intervention in this study.
* Any ongoing or recent (ie, during the screening period) minor medical complaints.
* Previous bone marrow transplant.
* Non leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Final Follow-up (FU) Visit (Week 10) or Early Termination (ET) (assessed up to 14 Weeks)
  To assess adverse events as a variable of safety and tolerability of AZD7503 following SC single dose administration.

SECONDARY OUTCOMES:
Area under plasma concentration time-curve from zero to infinity (AUCinf) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (AUCinf) of AZD7503 following SC administration of single ascending doses of AZD7503.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (AUClast) of AZD7503 following SC administration of single ascending doses of AZD7503.
Maximum observed plasma (peak) drug concentration (Cmax) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (Cmax) of AZD7503 following SC administration of single ascending doses of AZD7503.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (tmax) of AZD7503 following SC administration of single ascending doses of AZD7503.
Time of last observed (quantifiable) concentration (tlast) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (tlast) of AZD7503 following SC administration of single ascending doses of AZD7503.
Partial area under the plasma concentration-time curve from time 0 to time 48 hours post dose [AUC(0-48)] of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK [AUC(0-48)] of AZD7503 following SC administration of single ascending doses of AZD7503.
Half-life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (t½λz) of AZD7503 following SC administration of single ascending doses of AZD7503.
Mean residence time of the unchanged drug in the systemic circulation (MRTinf) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (MRTinf) of AZD7503 following SC administration of single ascending doses of AZD7503.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (CL/F) of AZD7503 following SC administration of single ascending doses of AZD7503.
Apparent volume of distribution at steady state following extravascular administration (Vz/F) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4 and final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To characterise the PK (Vz/F) of AZD7503 following SC administration of single ascending doses of AZD7503.
Cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4
  To characterise the PK [Ae(t1-t2)] of AZD7503 following SC administration of single ascending doses of AZD7503.
Percentage of dose excreted unchanged in urine from time t1 to t2 [Fe(t1-t2)] of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4
  To characterise the PK [Fe(t1-t2)] of AZD7503 following SC administration of single ascending doses of AZD7503.
Renal clearance of drug from plasma (CLR) of AZD7503 | (Pre-dose and Post-dose) Days 1 to 4
  To characterise the PK (CLR) of AZD7503 following SC administration of single ascending doses of AZD7503.
Number of participants with positive anti-drug antibodies (ADA) of AZD7503 | Day -1 to final FU visit (Week 10 post last dose) or ET (assessed up to 14 Weeks)
  To explore the formation of ADAs.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9230C00001&attachmentIdentifier=95cad428-bc71-48be-b805-dc7eff0b7ab5&fileName=D9230C00001_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search